CLINICAL TRIAL: NCT01594593
Title: Pilot Study of an Acceptance and Commitment Therapy Workshop for Distress and Decision Making in Early Stage Prostate Cancer in Veterans
Brief Title: Acceptance-Based Treatment for Prostate Cancer Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: Alliant International University (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 110353
Record Dates: First submitted 2012-04-23; First posted 2012-05-09 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Early Stage Prostate Cancer
Keywords: prostate cancer; behavioral; acceptance and commitment therapy; distress
MeSH Terms: conditions — Prostatic Neoplasms; Behavior | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental): Group-based behavioral workshop to address cancer-related distress
  Interventions: Behavioral: Acceptance and Commitment Therapy
- treatment as usual (No Intervention)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — group-based behavioral workshop to address cancer-related distress
  Arms: Acceptance and Commitment Therapy

SUMMARY:
Prostate cancer (PCa) is the most common type of cancer in men and the second leading cause of death in American men. Those diagnosed with localized prostate cancer encounter three sources of psychological distress: 1) diagnosis itself, 2) treatment decision making, and 3) the often life-altering side effects of treatment. In addition, patients who choose to undergo active surveillance which focuses on monitoring cancer in lieu of treatment, experience distress related to living with cancer. Acceptance and Commitment Therapy (ACT) is an established psychosocial intervention that has been used extensively for mental health treatment and has shown benefits for various chronic conditions. ACT is a behavioral intervention that focuses on tolerating distress and improving function. This pilot study is designed to test the feasibility of ACT for distress reduction and improved quality of life in patients recently diagnosed with early-stage, localized PCa.

ELIGIBILITY:
Inclusion Criteria:

* Localized prostate cancer in Stages I or II
* Ability to give informed consent
* Age 18 to 80 years old
* Willingness to come in for a day long intervention

Exclusion Criteria:

* Acute psychosis
* Suicidal ideation
* Homicidal ideation
* Active substance abuse
* Dementia

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of dropouts | 6 months
  Because this is a pilot study to determine feasibility, one of the primary outcomes is the number of participants who drop out of the active treatment arm.
Number of refusals | 6 months
  Because this is a pilot study to determine feasibility, one of the primary outcomes is the number of participants who refuse the active treatment arm.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | baseline, post intervention, 2 weeks post intervention, 3 months post intervention
Memorial Anxiety Scale for Prostate Cancer | baseline, post intervention, 2 weeks post intervention, 3 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Niloofar Afari, PhD, Principal Investigator — San Diego Veterans Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States